CLINICAL TRIAL: NCT04965038
Title: Early Reperfusion Therapy With Intravenous Thrombolysis for Recovery of VISION in Acute Central Retinal Artery Occlusion
Acronym: REVISION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-000183-29
Record Dates: First submitted 2021-06-15; First posted 2021-07-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-05

CONDITIONS: Central Retinal Artery Occlusion
Keywords: Central Retinal Artery Occlusion; Thrombolysis; Alteplase
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Thrombolysis (interventional study) (Active Comparator): Tenecteplase (0.25 mg per kg body weight as bolus; until trial protocol V04: Alteplase [0.9 mg per kg body weight; 10% as bolus; remaining over one hour] will be administered intravenously within 4.5 hours of symptom onset
  Interventions: Drug: Tenecteplase (until trial protocol V04: Alteplase)
- Placebo (interventional study) (Placebo Comparator): Placebo (0.25 mg per kg body weight as bolus; until trial protocol V04: 0.9 mg per kg body weight; 10% as bolus; remaining over one hour) will be administered intravenously within 4.5 hours of symptom onset
  Interventions: Drug: Tenecteplase (until trial protocol V04: Alteplase)
- Observational study (No Intervention): The prospective REVISION observational study will enroll patients within 12 hours of symptom onset

INTERVENTIONS:
Drug: Tenecteplase (until trial protocol V04: Alteplase) — Intravenous thrombolysis within 4.5 hours of symptom onset
  Arms: Placebo (interventional study); Thrombolysis (interventional study)

SUMMARY:
Non-arteritic, thromboembolic central retinal artery occlusion (CRAO) is an acute neurovascular-ophthalmological emergency which leads to severe and permanent vision loss; no evidence-based therapy does exist. Two recent meta-analyses indicate early intravenous thrombolysis to be beneficial in CRAO. Therefore, the REVISION randomized placebo-controlled interventional trial will investigate intravenous alteplase in CRAO as it is practiced in acute ischemic stroke, i.e. within 4.5 hours after symptom onset.

The REVISION observational study will evaluate retinal changes on optical coherence tomography (OCT) in patients within 12 hours of CRAO onset, and the REVISION substudy, which will be conducted adjunct to either the interventional or the observational study, will evaluate the value of the retrobulbar spot sign for prediction of outcome and treatment response.

DETAILED DESCRIPTION:
Non-arteritic, thromboembolic central retinal artery occlusion (CRAO) is an acute neurovascular-ophthalmological emergency which leads to severe and permanent vision loss in the affected eye in ~ 95% of cases. Despite a variety of widely practiced "conservative standard treatments", such as hemodilution, ocular massage, and paracentesis, there is no evidence-based therapy for non-arteritic CRAO. Animal models have proven a limited ischemic tolerance of the retina with irreversible damage occurring within only four hours after disruption of blood flow. This is why rapid reperfusion represents THE logical therapeutic approach. Two recent meta-analyses indicate early intravenous thrombolysis to be beneficial in CRAO. Therefore, the REVISION trial will investigate intravenous alteplase in CRAO as it is practiced in acute ischemic stroke, i.e. within 4.5 hours after symptom onset.

Sequential evaluation by optical coherence tomography (OCT) will visualize dynamic ischemic changes of the retina during and after CRAO. The REVISION observational study will enroll patients within 12 hours of symptom onset and aims at comparing late time window retinal findings to early ischemic changes found in patients of the randomized REVISION interventional trial. Ultimately, OCT may become the preferred tool when it comes to assess retinal tissue viability in patients with an unknown CRAO onset (e.g. wake-up CRAO), and CRAO patients who present in an extended time window beyond 4.5 hours.

The REVISION substudy, which will be conducted adjunct to either the interventional or the observational study, will evaluate the value of the retrobulbar spot sign for prediction of outcome and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Acute non-arteritic CRAO (i.e. sudden, painless monocular vision loss) ≤ 12 hours after symptom onset confirmed by an experienced ophthalmologist through assessment of: BCVA, intraocular pressure, swinging flash light test (relative afferent pupil defect), slit-lamp biomicroscopy, fundoscopy, and OCT of the macula of both eyes* (*within the 4.5-hour time window: to be skipped if not feasible ≤ 10 minutes; beyond the 4.5-hour time window: mandatory)
* BCVA of LogMAR ≥ 1.3 in the affected eye (functional blindness according to WHO ICD-11)
* Reading must have been possible with the affected eye before CRAO (LogMAR ≤ 0.5)
* Neurological examination performed by an experienced stroke neurologist
* Brain imaging as per local standard for acute retinal ischemia/stroke assessment, either cranial computed tomography (CT) or cranial magnetic resonance imaging (MRI)

Exclusion Criteria:

* Suspected giant cell arteritis
* Other-than-CRAO cause of acute visual loss (e.g., retinal detachment, vitreous hemorrhage, acute glaucoma, acute optic neuritis)
* BCVA of LogMAR < 1.3 or rapidly improving vision in the affected eye
* Acute ischemic stroke with indication for on-label intravenous thrombolysis (IVT)
* Any co-existing or terminal disease with anticipated life expectancy of < 3 months
* Prior participation in the REVISION trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery at visit 3 | 30 days
  Functional recovery to best corrected visual acuity of logarithm of the minimum angle of resolution ≤ 0.5 in the affected eye, which corresponds to normal to mild vision impairment (intention-to-treat analysis).

SECONDARY OUTCOMES:
best corrected visual acuity (BCVA) at visits 2, 3, and 4 | 90 days
  Functional recovery to best corrected visual acuity of logarithm of the minimum angle of resolution ≤ 0.5 in the affected eye, which corresponds to normal to mild vision impairment (intention-to-treat and per-protocol analyses).
Shift in visual outcome categories at visits 2, 3, and 4 | 90 days
  Shift in visual outcome categories: normal vision (logarithm of the minimum angle of resolution (LogMAR) ≤ 0), mild vision impairment (LogMAR > 0 and ≤ 0.5), moderate vision impairment (LogMAR > 0.5 and ≤ 1.0), severe vision impairment (LogMAR > 1.0 and ≤ 1.3), counting fingers (LogMAR > 1.3 and ≤ counting fingers), hand motion or light perception, and no light perception.
Dichotomized analysis of visual outcome at visits 2, 3, and 4 | 90 days
  Dichotomized analysis of visual outcome: 'normal vision to moderate vision impairment' vs. 'severe vision impairment or functional blindness' and 'normal vision to severe vision impairment' vs. 'functional blindness'.
Visual field at visits 3 and 4 | 90 days
  Kinetic visual field using III4e mark
Central retinal artery recanalization at visits 2, 3, and 4 | 90 days
  Central retinal artery recanalization assessed using optical coherence tomography angiography (OCTA) of the optic nerve head and the macula.
Retinal arterial perfusion at visits 3 and 4 | 90 days
  Retinal arterial perfusion assessed using fluorescein angiography.
National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) at visits 3 and 4 | 90 days
  NEI-VFQ-25 for assessment of relevant visual impairment
National Institutes of Health Stroke Scale (NIHSS) score at visit 2 | 72 hours
  NIHSS for assessment of neurological deficits due to ischemic stroke or intracranial hemorrhage
Modified Rankin Scale (mRS) score at visits 3 and 4 | 90 days
  Dichotomized analysis and shift analyses of mRS (categories 0 - 1 (excellent outcome) vs. 2 - 6, 0 - 2 (functional independence) vs. 3 - 6, 0 - 3 (walking) vs. 4 - 6, and 0 - 4 vs. 5 - 6 (bedridden or death), and shift analysis)
Fresh ischemic lesions on cranial magnetic resonance imaging (MRI) at visit 2 | 72 hours
  Fraction of patients with and number of acute ischemic lesions on follow-up diffusion-weighted cranial MRI
Death at visits 3 and 4 | 90 days
  All-cause and stroke-related death
Any intracranial hemorrhage (ICH) at visit 2 | 72 hours
  Any ICH (except microhemorrhages) on follow-up magnetic resonance imaging; in case of missing follow-up brain imaging due to premature death, ICH will be replaced by "ICH or death without repeat scan")
Symptomatic intracranial hemorrhage (ICH) until visit 2 | 72 hours
  Symptomatic ICH (as per ECASS III and Heidelberg bleeding classification) until follow-up magnetic resonance imaging; in case of missing follow-up brain imaging due to premature death, symptomatic ICH will be replaced by "symptomatic ICH or death without repeat scan")
Intraocular hemorrhage in the affected eye at visit 2 | 72 hours
  Intraocular hemorrhage in the affected eye
Major bleeding until visit 2 | 72 hours
  Major bleeding, defined as clinically overt bleeding associated with at least one of the following features: decrease in hemoglobin levels of ≥ 2 g/dL over 24 hours, bleeding requiring transfusion of ≥ 2 units of packed red cells, bleeding at a critical site (i.e., intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, or retroperitoneal), or bleeding resulting in the death of the patient
Retinal neovascularization requiring therapy at visit 3 and 4 | 90 days
  Retinal neovascularization requiring therapy
(Serious) adverse events ((S)AE) | 90 days
  AE until visit 2, serious AE and AE of special interest until visit 3 and 4

OTHER OUTCOMES:
Exploratory Outcomes of the REVISION Interventional Study | 90 days
  Optical coherence tomography/angiography (OCT/A) findings at screening, visit 2, 3, and 4 as prognostic biomarkers for prediction of time since CRAO onset, visual outcomes, and treatment response; to identify respective thresholds which are incompatible with a satisfactory IVT response and/or functional recovery
Exploratory Outcomes of the REVISION Observational Study | 1 day
  Optical coherence tomography/angiography (OCT/A) findings at screening as prognostic biomarker for prediction of time since CRAO onset and visual outcomes, and to compare extended time window results to those of interventional study participants.
Exploratory Outcomes of the Retrobulbar Spot Sign Substudy | 30 days
  To investigate the retrobular spot sign on transorbital ultrasound at visits 2 and 3 as prognostic biomarker for prediction of treatment response and visual outcomes; to compare central retinal artery recanalization assessment with transorbital ultrasound with that using optical coherence tomography/angiography (OCT/A) of the optic nerve head and the macula, and fluorescein angiography

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poli S, Grohmann C, Wenzel DA, Poli K, Tunnerhoff J, Nedelmann M, Fiehler J, Burghaus I, Lehmann M, Glauch M, Schadwinkel HM, Kalmbach P, Zeller J, Peters T, Eschenfelder C, Agostini H, Campbell BC, Fischer MD, Sykora M, Mac Grory B, Feltgen N, Kowarik M, Seiffge D, Strbian D, Albrecht M, Alzureiqi MS, Auffarth G, Bazner H, Behnke S, Berberich A, Bode F, Bohmann FO, Cheng B, Czihal M, Danyel LA, Dimopoulos S, Pinhal Ferreira de Pinho JD, Fries FN, Gamulescu MA, Gekeler F, Gomez-Exposito A, Gumbinger C, Guthoff R, Hattenbach LO, Kellert L, Khoramnia R, Kohnen T, Kurten D, Lackner B, Laible M, Lee JI, Leithner C, Liegl R, Lochner P, Mackert M, Mbroh J, Muller S, Nagel S, Prasuhn M, Purrucker J, Reich A, Mundiyanapurath S, Royl G, Salchow DJ, Schafer JH, Schlachetzki F, Schmack I, Thomalla G, Tieck Fernandez MP, Wakili P, Walter P, Wolf A, Wolf M, Bartz-Schmidt KU, Schultheiss M, Spitzer MS. Early REperfusion therapy with intravenous alteplase for recovery of VISION in acute central retinal artery occlusion (REVISION): Study protocol of a phase III trial. Int J Stroke. 2024 Aug;19(7):823-829. doi: 10.1177/17474930241248516. Epub 2024 Jun 25. PMID 38591748